CLINICAL TRIAL: NCT05273853
Title: Speech Outcome After Partial Adenoidectomy in Patients With Risk of Hypernasality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Dina Awida Hasb Allah, Resident of Otolaryngology, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DAHAllah
Record Dates: First submitted 2022-02-18; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Hypernasality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with high risk of hypernasality (Other): In 1958, Gibb indicated an incidence of hypernasality (escape of air from nose as in patients with cleft palate) postadenoidectomy in approximately 1of 2000 cases. Closure pattern of velopharyngeal valve in children is veloadenoidal rather than velopharyngeal closure. Adenoid tissue is vital to velopharyngeal closure in children and its removal necessitates a change in the closure pattern of velopharyngeal valving. These changes are easily overcome if there is no anatomic abnormality
  Interventions: Procedure: Partial Adenoidectomy

INTERVENTIONS:
Procedure: Partial Adenoidectomy — Partial removal of adenoid

SUMMARY:
Adenoid hypertrophy is a common cause of airway obstruction in children; it may lead to mouth breathing, nasal discharge, snoring, sleep apnea, and hyponasal speech.

DETAILED DESCRIPTION:
Adenoid hypertrophy is a common cause of airway obstruction in children; it may lead to mouth breathing, nasal discharge, snoring, sleep apnea, and hyponasal speech. It also contributes to the pathogenesis of rhinosinusitis and recurrent otitis media. However, the adenoid lies in the posterior nasopharyngeal wall and may act as a pad against the palate facilitating velopharyngeal closure, especially in patients with palatal abnormalities; Its presence can compensate for a short or poorly mobile palate. Following adenoidectomy, compensation is eliminated and velopharyngeal insufficiency (VPI) may result. Therefore, patients with palatal abnormalities (such as poor palatal mobility, short palate, occult submucosal cleft palate, scarred palate after previous tonsillectomy, and repaired cleft palate) are at high risk to develop hypernasality after complete adenoidectomy, and in such situations conservative or partial adenoidectomy is performed

ELIGIBILITY:
Inclusion Criteria:

1. Patient with symptoms of adenoid hypertrophy.
2. High risk to VPI:

   1. Short palate.
   2. Scarred palate after previous tonsillectomy.
   3. Occult submucous cleft.
   4. Deep pharynx.
   5. Repaired cleft palate.

Exclusion Criteria:

* Any neurological deficit, muscular disorder or structural defects of the palate (as cleft palate).

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-08-04 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Speech Outcome | 1 month after operation
  Change of a degree of Nasal Tone during speech
Speech Outcome | 3 months after operation
  Change of a degree of Nasal Tone during speech

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed AE Ahmed, Professor, Study Chair — Sohag Faculty Of Medicine
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rowe MR, D'Antonio LL. Velopharyngeal dysfunction: evolving developments in evaluation. Curr Opin Otolaryngol Head Neck Surg. 2005 Dec;13(6):366-70. doi: 10.1097/01.moo.0000186204.53214.62. PMID 16282766